CLINICAL TRIAL: NCT00992719
Title: A Phase II Study In Pregnant Women to Assess the Safety and Immunogenicity of an Unadjuvanted Novartis H1N1 Inactivated Influenza Vaccine Administered at Two Dose Levels
Brief Title: Novartis H1N1 Vaccine in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0072; N01AI80057C
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2012-03-05 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2010-07

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, pregnant women
MeSH Terms: conditions — Influenza, Human

ARMS (3):
- Group 3: Non-pregnant Women: 15 mcg H1N1 Vaccine (Active Comparator): 100 non-pregnant women to receive 15 mcg inactivated H1N1 vaccine.
  Interventions: Biological: Inactivated H1N1 Vaccine
- Group 2: Pregnant Women: 30 mcg H1N1 Vaccine (Experimental): 100 pregnant women to receive 30 mcg inactivated H1N1 vaccine.
  Interventions: Biological: Inactivated H1N1 Vaccine
- Group 1: Pregnant Women: 15 mcg H1N1 Vaccine (Experimental): 100 pregnant women to receive 15 mcg inactivated H1N1 vaccine.
  Interventions: Biological: Inactivated H1N1 Vaccine

INTERVENTIONS:
Biological: Inactivated H1N1 Vaccine — H1N1 vaccine [Influenza A (H1N1) 2009 Monovalent Vaccine] is a licensed, inactivated influenza virus vaccine. It will be provided as prefilled single dose syringes containing 0.5 mL. The 0.5 mL prefilled syringe is formulated without preservative. The 15 microgram (mcg) dose will be administered as a single 0.5 mL intramuscular (IM) injection in the deltoid muscle of the preferred arm. The 30 mcg dose will be administered as two 0.5 mL injections in the deltoid muscle of each arm.

SUMMARY:
The purpose of this study is to evaluate the safety of a 2009 H1N1 influenza vaccine in pregnant women and to determine how their body reacts to different strengths of the vaccine. Two strengths of the H1N1 influenza vaccine will be tested. Since it is not known if the response to the vaccine in pregnant women is the same or different than in non-pregnant women, the study also includes a group of women who are not pregnant for comparison. Participants include 200 pregnant women and 100 non-pregnant women ages 18-39. Study procedures include physical exams, several blood samples and maintaining a memory aid to document daily temperature and side effects for 8 days following vaccination. Participants will be involved in study related procedures for about 6 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization to declare a pandemic on June 11, 2009. Pregnant women are at an increased risk for serious consequences of influenza infection. A 15 microgram (mcg) dose of unadjuvanted inactivated H1N1 vaccine is recommended for healthy adults and recent preliminary data indicates this dose is likely to be protective for pregnant women. However, a higher dose of an unadjuvanted, inactivated influenza H1N1 vaccine may be necessary to confer optimal protection to this at risk population. This protocol will explore the antibody response following vaccination of pregnant women at 2 different dose levels (15 mcg and 30 mcg) and a non-pregnant control group receiving a 15 mcg dose. Antibody responses will be assessed at 21 days and 180 days post vaccination. For pregnant women, maternal and cord blood will be collected to determine the level of H1N1 antibodies transferred to the baby. An optimal immune response in pregnant women would impact transplacental transport of protective antibodies which is important since vaccines are not available for infants younger than six months, another at risk population for severe H1N1 disease. Sustained immunity for at least 6 months post-vaccination would impart benefit not only to the woman herself but also decrease a primary exposure risk (infected mother) for the newborn infant. Furthermore, a systematic evaluation of the kinetics of maternally transferred antibodies to 2009 H1N1 influenza virus will help improve and develop strategies to protect infants from influenza. This is an open label, Phase II study in pregnant and non-pregnant women, aged 18-39 years old designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine. Pregnant women will be randomized into 2 groups (100 per dose group) to receive intramuscular (IM) inactivated influenza H1N1 vaccine at 15 mcg (Group 1) or 30 mcg (Group 2). A non-pregnant control group of 100 subjects will receive IM inactivated influenza H1N1 vaccine at 15 mcg (Group 3). Following immunization, safety will be measured by assessment of adverse events (AEs) through 21 days post vaccination (serious AEs and new-onset chronic medical conditions monthly through 6 months post vaccination (Day 180). Reactogenicity to the vaccine will be assessed for 8 days following vaccination (Day 0-7). Immunogenicity testing will include hemagglutination inhibition assay (HAI) and neutralizing antibody testing on serum obtained on Days 0, 21, and 180. For the pregnant groups, HAI antibody testing will also be performed on serum from the participant at delivery, on serum from cord blood collected at delivery and, when possible, on serum samples collected from the participant at day 180 and from the infant at 6 weeks, four months, or six months after delivery. The primary safety objective is to assess the safety of unadjuvanted, inactivated H1N1 influenza vaccine in pregnant women when administered at the 15 mcg or 30 mcg dose. The primary immunogenicity objective is to assess the antibody response to unadjuvanted, inactivated H1N1 influenza vaccine in pregnant women when administered at the 15 mcg or 30 mcg dose. The secondary objective for pregnant women is to assess the efficiency of placental transport of maternal influenza antigen specific antibodies to the neonate.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

* Pregnant female between the ages of 18 and 39 years, inclusive.
* Is from 14 weeks/0 days through 33 weeks/6 days of gestation.
* Had at least one prenatal visit during which pregnancy was confirmed.
* Is in good health, as determined by vital signs (heart rate less than or equal to 100 beats per minute; blood pressure: systolic less than or equal to 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature less than or equal to 100 degrees Fahrenheit), medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history.
* Receipt of the 2009-2010 seasonal influenza vaccine no less than two weeks prior to enrollment in this study.
* Intend to be available through 6 months following receipt of H1N1 vaccine.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.
* Agrees to sign medical release for herself and her infant(s) to allow study staff to gather pregnancy outcome data, if needed per clinical site policy.

Non-pregnant women:

* Female between the ages of 18-39 years, inclusive.
* For the 30 days prior to enrollment through 30 days following receipt of H1N1 vaccine must fulfill one of the following: (i) she is not able to bear children because she has been surgically sterilized (tubal ligation or hysterectomy) for at least one year or is at least 1 year post-menopausal or (ii) she agrees to practice effective methods of contraception including, but not limited to, abstinence, barrier methods (such as a condom or diaphragm) used with a spermicide, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices).
* For a female subject of childbearing potential, must have a negative pregnancy test (urine or serum) within 24 hours prior to vaccination.
* Is in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history (if indicated). A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
* Receipt of the 2009-2010 seasonal influenza vaccine no less than two weeks prior to enrollment in this study
* Intend to be available for a follow-up visit and phone call access through 6 months following receipt of H1N1 vaccine.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

Pregnant women:

* Has a known allergy or hypersensitivity to eggs or other components in the vaccines (these may include, but are not limited to: polymyxin and neomycin).
* Has a history of severe reactions following previous immunization with influenza virus vaccines.
* Has participated in a novel influenza H1N1 2009 vaccine study in the past 2 years, has received a H1N1 2009 vaccine or has history of novel influenza H1N1 2009 infection evaluated by a healthcare professional prior to enrollment.
* Has received any other live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following vaccination. Measles, mumps, and rubella vaccine and tetanus, diphtheria, and acellular pertussis vaccine and human papillomavirus vaccine are permitted post-partum.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expects to receive another experimental/investigational agent during the study period (prior to 180 days post vaccination).
* Has an acute illness and/or an oral temperature >/= 100.0 F, within 72 hours of vaccination (This may result in a temporary delay of vaccination).
* Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants.
* Long term use of glucocorticoids, including oral or parenteral, or high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed) or has received betamethasone or dexamethasone to accelerate fetal lung maturity.
* Has a history of receiving immunoglobulin or other blood product (with exception of Rhogam) within the 3 months prior to enrollment in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* The subject is receiving any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving an antidepressant drug (not listed above) and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of alcohol or drug abuse in the last 5 years.
* Has a seizure disorder or is on an anti-seizure medication.
* Has a history of Guillain-Barré Syndrome.
* Plan to travel outside of North America in the time between vaccination and 21 days following vaccination
* Has an acute or chronic medical condition that, in the opinion of the investigator would render vaccination unsafe, or would interfere with the evaluation of responses (this includes, but is not limited to, known cardiac disease, chronic liver disease, significant renal disease, unstable or progressive neurological disorder, transplant recipients or uncontrolled diabetes, juvenile diabetes (Type I) or advanced diabetes with renal disease or eye disease, diabetes controlled by diet or insulin is acceptable).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Non-pregnant women:

* Has a known allergy or hypersensitivity to eggs, egg proteins, other components in the vaccines (these may include, but not limited to: polymyxin and neomycin).
* Has a history of severe reactions following previous immunization with influenza virus vaccines.
* Has participated in a novel influenza H1N1 2009 vaccine study in the past 2 years, has received H1N1 2009 vaccine or has history of novel influenza H1N1 2009 infection evaluated by a healthcare professional prior to enrollment.
* Has received any other live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following vaccination.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expects to receive another experimental/investigational agent during the study period (prior to 180 days post vaccination).
* Is breastfeeding or intends to become pregnant during the study period between enrollment and 30 days following receipt of the H1N1 vaccine.
* Has an acute illness and/or an oral temperature greater than or equal to 100.0 F, within 72 hours of vaccination (This may result in a temporary delay of vaccination).
* Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants.
* Long term use of glucocorticoids, including oral or parenteral, or high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* The subject is receiving any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving an antidepressant drug (not listed above) and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* History of alcohol or drug abuse in the last 5 years.
* Has a seizure disorder or is on an anti-seizure medication.
* Has a history of Guillain-Barré Syndrome.
* Plan to travel outside of North America in the time between vaccination and 21 days following vaccination.
* Has an acute or chronic medical condition that, in the opinion of the investigator would render vaccination unsafe, or would interfere with the evaluation of responses (this includes, but is not limited to, known cardiac disease, chronic liver disease, significant renal disease, unstable or progressive neurological disorder, transplant recipients or uncontrolled diabetes, juvenile diabetes (Type I) or advanced diabetes with renal disease or eye disease, diabetes controlled by diet or insulin is acceptable.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine - Department of Molecular Virology and Microbiology, Houston, Texas
  - Group Health Cooperative, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy pregnant and non-pregnant women recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 09Nov2009 and 04May2010.
Groups:
- Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine: Pregnant participants received 15 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0
- Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine: Pregnant participants received 30 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0
- Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine: Non-pregnant participants received 15 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0
Period: Overall Study
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Started | 28 | 28 | 28
Completed | 27 | 27 | 28
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine | Total
Number analyzed (Participants) | 28 | 28 | 28 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 28 | 84
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (6.0) | 28.8 (4.9) | 30.8 (5.6) | 29.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 28 | 84
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 28 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Maternal Complications of Pregnancy, Labor and Delivery
Description: Participants were contacted after delivery, and medical records reviewed, to collect complications experienced during pregnancy, labor and delivery. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery
Population: All participants from whom outcome data were collected are included in the ITT safety population for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 27 | 28
participants
  Stillborn | 0 | 0
  Miscarriage | 0 | 0
  Gestational diabetes | 1 | 2
  Polyhydramnios | 1 | 0
  Oligohydramnios | 1 | 1
  Pregnancy induced hypertension | 0 | 3
  Pre-eclampsia | 1 | 3
  Eclampsia | 0 | 0
  Fetal Distress | 2 | 1
  Abruptio Placenta | 0 | 1
  Chorioamnionitis | 0 | 0
  Fever | 2 | 1
  Anaphylaxis | 0 | 0
  Antibiotics prior to delivery | 12 | 12
  Fetal abnormalities detected during pregnancy | 1 | 0
  Assisted vaginal delivery | 1 | 1
  Non-elective Cesarean section | 6 | 3
  Abnormal amniotic fluid | 5 | 5
  Postpartum fever | 0 | 0
  Postpartum endometritis | 0 | 0
  Postpartum bleeding | 2 | 0
  Postpartum bacteremia | 0 | 0

2. Primary Outcome: Number of Births With Neonatal Complications
Description: Participants were contacted after delivery, and medical records reviewed, to collect neonatal complications. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery
Population: All births are included in this outcome measure. Two participants gave birth to twins and two to triplets, each counted separately.
Measure: Number; unit: births
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 29 | 32
births
  Pre-term (less than 37 weeks) | 5 | 9
  Large for gestational age | 6 | 2
  Small for gestational age | 0 | 3
  Abnormal infant exam | 1 | 4
  Congenital abnormalities | 0 | 1
  Hematological complications | 1 | 1
  Infections | 0 | 0
  Sepsis | 0 | 0
  Meningitis | 0 | 0
  Metabolic complications | 1 | 1
  Respiratory complications | 5 | 4
  Respiratory support used | 5 | 4
  Fever 100.4 degrees Fahrenheit or greater | 0 | 0
  Admission to special nursery/infant intensive care | 5 | 8

3. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death of the mother, fetus or infant; was life threatening to mother, fetus or infant; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; was a congenital anomaly/birth defect in fetus or infant; or may have jeopardized the mother, fetus or infant, or required intervention to prevent one of the outcomes, or was described as Guillain-Barré Syndrome. Association was determined by a clinician licensed to diagnose and listed on the site's FDA Form 1572.
Time Frame: Day 0 through Day 180 after vaccination
Population: All participants receiving the vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 28 | 28 | 28
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days post vaccination (Day 0-7)
Population: All participants receiving the vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 28 | 28 | 28
participants
  Pain | 4 | 8 | 6
  Tenderness | 13 | 15 | 14
  Swelling | 1 | 2 | 2

5. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Within 8 days post vaccination (Day 0-7)
Population: All participants receiving the vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 28 | 28 | 28
participants
  Redness | 2 | 2 | 2
  Swelling | 1 | 1 | 2

6. Secondary Outcome: Number of Participants With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer Greater Than or Equal to 40 Against the Novel Influenza H1N1 2009 Virus in the Maternal Blood at the Time of Delivery
Description: Blood was collected from participants at the time of delivery for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: At time of delivery
Population: Pregnant participants were included in the analyses if they had blood collected at delivery, with 1 participant excluded due to receipt of non-study vaccine. Participants were analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 25 | 22
participants | 17 | 16

7. Secondary Outcome: Number of Participants With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer Greater Than or Equal to 40 Against the Novel Influenza H1N1 2009 Virus in Cord Blood
Description: Cord blood was collected at the time of delivery for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: At time of delivery
Population: Pregnant participants were included in the analyses if they had cord blood collected at delivery, with 1 participant excluded due to receipt of non-study vaccine. Participants were analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 22 | 22
participants | 17 | 18

8. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days post vaccination (Day 0-7)
Population: All participants receiving the vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 28 | 28 | 28
participants
  Feverishness | 0 | 2 | 3
  Malaise | 7 | 14 | 4
  Myalgia | 1 | 6 | 4
  Headache | 8 | 9 | 7
  Nausea | 3 | 8 | 3

9. Primary Outcome: Number of Participants Reporting Fever After Vaccination
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 37.8 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 37.8 degrees Celsius or higher on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post vaccination
Population: All participants receiving the vaccination and who reported temperatures are included in the safety cohort. One participant did not report temperatures. Analyses are as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 28 | 27 | 28
participants | 1 | 0 | 0

10. Primary Outcome: Number of Participants With 4-fold or Greater Serum Hemagglutination Inhibition (HAI) Antibody Titer Increases Against Influenza H1N1 2009 Virus Following a Single Dose of H1N1 Vaccine
Description: Blood was collected from all participants prior to vaccination as well as 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 21 after the first vaccination
Population: Participants were included in the analyses if they received the vaccination and had blood collected at both timepoints, with 1 participant excluded due to receipt of non-study vaccines. Participants were analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 26 | 28 | 28
participants | 18 | 26 | 24

11. Primary Outcome: Number of Participants With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus Following a Single Dose of H1N1 Vaccine
Description: Blood was collected from all participants prior to and at Day 21 post vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0 prior to and Day 21 following vaccination
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Number analyzed (Participants) | 26 | 28 | 28
participants
  Day 0 | 5 | 3 | 2
  Day 21 | 22 | 27 | 26

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after vaccination, unsolicited events through 21 days after vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after vaccination, including at the time of delivery.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 8/28 | 6/28 | 1/28
Other Adverse Events (participants affected / at risk) | 19/28 | 24/28 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine (N=28) | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine (N=28) | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine (N=28)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 0 (0)
Amniorrhoea (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (2) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Pregnant Women: 15 Mcg H1N1 Vaccine (N=28) | Group 2: Pregnant Women: 30 Mcg H1N1 Vaccine (N=28) | Group 3: Non-pregnant Women: 15 Mcg H1N1 Vaccine (N=28)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 6 (6)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 3 (3)
Malaise (General disorders) | 7 (7) | 14 (14) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 9 (9) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (8) | 3 (3)
Injection site pain (General disorders) | 4 (4) | 8 (8) | 6 (6)
Tenderness (General disorders) | 13 (13) | 15 (15) | 14 (14) — Solicited as a reaction at the vaccination site
Injection site erythema (General disorders) | 2 (2) | 2 (2) | 2 (2)
Injection site swelling (functional grading) (General disorders) | 1 (1) | 2 (2) | 2 (2) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 1 (1) | 1 (1) | 2 (2) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

LIMITATIONS AND CAVEATS:
Although 200 pregnant and 100 non-pregnant subjects were targeted for enrollment, enrollment closed in May 2010 prior to reaching the target due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less